CLINICAL TRIAL: NCT02658864
Title: Pharmacokinetic Properties and Effect of Food on Pharmacokinetic Properties of the Oral Lafutidine Tablets in Healthy Chinese Subjects
Brief Title: Pharmacokinetic Properties and Effect of Food on Pharmacokinetic Properties of the Oral Lafutidine Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Weiyong Li, vice director of the pharmcy department, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: WHXH-lafutidine
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Gastritis
Keywords: lafutidine tablet; pharmacokinetics; food; safety; healthy subjects
MeSH Terms: interventions — lafutidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 10-mg group (Experimental): Twelve healthy subjects were administered a single oral dose of 10 mg lafutidine tablets in fasted state.
  Interventions: Drug: lafutidine
- 20-mg group (Experimental): Twelve healthy subjects were administered a single oral dose of 20 mg lafutidine tablets in fasted state.
  Interventions: Drug: lafutidine
- 40-mg group (Experimental): Twelve healthy subjects were administered a single oral dose of 40 mg lafutidine tablets in fasted state.
  Interventions: Drug: lafutidine

INTERVENTIONS:
Drug: lafutidine — comparison of different doses, sex and medication conditions

SUMMARY:
This study was to evaluate the pharmacokinetics of single and multiple doses of oral lafutidine tablets and the effect of food on pharmacokinetics in healthy Chinese subjects. The tolerability and the effect of sex on the pharmacokinetic properties were also evaluated to acquire more pharmacokinetic information.

DETAILED DESCRIPTION:
The study of single-dose was randomized, three-period, crossover. And in this study, 12 subjects were randomly assigned to 3 dose groups and received a single dose of 10mg, 20mg and 40mg lafutidine tablets. The washout period was 7 calendar days. In the multiple-dose, 12 subjects took lafutidine tablets of 10 mg twice a day for 6 consecutive days. In the food-effect study, 12 subjects were randomly assigned to 2 groups. One group received a single dose of 10mg lafutidine tablets under fasted condition, while the other were in fed condition. The drug administrations were separated by a wash-out period of seven calendar days. In each study group, the male and the female are both in half of the subjects. Using a liquid chromatography tandem mass spectrometry (LC/MS/MS) method to determine the plasma concentration of lafutidine. Pharmacokinetic parameters were calculated using the single compartment model.

ELIGIBILITY:
Inclusion Criteria:

* body mass index between19 and 24 kg/m2
* negative for HIV and hepatitis B
* had no clinical important findings on health tests
* thorax radiography and ECG with no abnormalities
* normal blood pressure values
* heart rate

Exclusion Criteria:

* any drug treatment within 2 weeks before starting the study
* participation in another clinical study within the previous 3 months
* alcoholism and smoking
* pregnancy
* breast-feeding
* hypocalcemia
* blood donation or participation in other clinical trials within 3 months before enrollment in the study
* sitting blood pressure <80/50 mm Hg or >140/100 mm Hg
* A ventricular rate <60 beats/min or >100 beats/min at rest

Ages: 19 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2005-04; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Cmax | one day
  Peak concentration
Area under the curve | one day
  Area under the curve - plasma concentration
Clearance | one day
  Clearance
Apparent volume of distribution-V | one day
  The apparent volume of distribution

SECONDARY OUTCOMES:
Safety (adverse events) | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Weiyong Li, PhD, Principal Investigator — HUST/Union Hospital